CLINICAL TRIAL: NCT01887483
Title: A Double-Blind Placebo-Controlled Randomized Clinical Trial Assessing the Effect of 2 Month Consumption of Vetal Laban Including L. Acidophilus on Functional Gastrointestinal Symptoms Among Subjects Fulfilling Rome III Criteria for IBS
Brief Title: Vetal Laban Intervention Trial Assessing Bowel Symptoms
Acronym: KF_2013
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow recruitment, high drop-out
Sponsor: Danisco (Industry)
Collaborators: Almarai (Unknown); Clinart International (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: KF_2013
Record Dates: First submitted 2013-05-27; First posted 2013-06-27 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2015-12

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS; bowel function; probiotic
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Lacteol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vetal Laban active (Active Comparator): Vetal Laban with L. acidophilus
  Interventions: Dietary Supplement: Vetal Laban active
- Placebo (Placebo Comparator): Vetal Laban -like product without L. acidophilus
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Vetal Laban active — Dairy product with probiotic
  Other Names: Vetal Laban, Lactobacillus acidophilus
  Arms: Vetal Laban active
Dietary Supplement: Placebo — Dairy product without probiotic
  Other Names: Vetal Laban-like product without L. acidophilus
  Arms: Placebo

SUMMARY:
A two month intervention trial assessing the effect of Vetal Laban containing L. acidophilus on enhancing functional bowel wellbeing among subjects with irritable bowel syndrome (IBS).

ELIGIBILITY:
Inclusion Criteria:

* Males and females aged 18 to 65 years
* Subjects fulfilling Rome III criteria for IBS
* Sufficient health and orientation for participating in the trial
* Obtained his/her informed consent after verbal and written information.
* Have a high probability for compliance with and completion of the study.
* Body Mass Index (BMI) between 19 and 35.

Exclusion Criteria:

* Diagnosed or suspected organic gastrointestinal disease (i.e. colitis, Crohn's disease, celiac disease, major bowel surgery, recurrent diverticulitis) or severely impaired general health including cancer and cancer therapy.
* Lactose intolerance
* Unwillingness to refrain from probiotic use during the trial
* Use of antibiotics within the 3 preceding months prior to recruitment
* Pregnant, planning pregnancy or lactating
* Expected major lifestyle changes related to nutrition, exercise, travelling etc.
* Participation in a clinical trial with an investigational product or drug within 3 months prior to screening.
* Substance abuse
* Subjects unable to read and understand the questionnaires

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
change in functional bowel symptoms | week 0, 4, 8, 12 and 16
  Validated questionnaire

SECONDARY OUTCOMES:
change in adequate relief of bowel symptoms | weekly from week 4 to week 12
  Weekly question
change in stool defecation frequency | week 0, 4, 8, 12 and 16
  Validated scale
change in stool microbiota | week 4, 8, 12 and 16
  molecular analyses
change in prevalence of adverse events | continuous from week 0 to 16
  Recording of adverse and serious adverse events
change in stool consistency | week 0, 4, 8, 12 and 16
  Validated scale

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Aljahdali, MD, Principal Investigator — King Abdulaziz National Guard Hospital, Riyadh, Kingdom of Saudi Arabia; Arthur C Ouwehand, PhD, Study Chair — Danisco Sweeteners Ltd.; Anna H Lyra, PhD, Study Director — Danisco Sweeteners Ltd.; Suzanne Alodaib, MSc, Study Director — Almarai Company, Saudi Arabia; Abed Allehibi, Dr, Principal Investigator — King Fahd Medical City; Othman Al-Harbi, Dr, Principal Investigator — King Khalid University Hospital
Locations (2):
- Saudi Arabia (2):
  - King Fahd Medical City, Riyadh
  - King Khalid University Hospital, Riyadh